CLINICAL TRIAL: NCT05383521
Title: Oral Tinidazole Treatment of Refractory Trichomonas Vaginitis
Brief Title: Safety and Efficacy of Two Oral Tinidazole Regimens for Refractory Trichomonas Vaginitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shangrong Fan (Other)
Responsible Party: Sponsor-Investigator, Shangrong Fan, Profesor, Peking University Shenzhen Hospital
Organization: Peking University Shenzhen Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020PUSZH001
Record Dates: First submitted 2021-01-05; First posted 2022-05-20 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Trichomonas Vaginitis
Keywords: Refractory Trichomonas Vaginitis; Tinidazole
MeSH Terms: conditions — Trichomonas Vaginitis

STUDY DESIGN:
Intervention Model Description: For patients who failed to conventional treatment (recommended by the guidelines including tinidazole, 2g once daily for 5-7 days), the following regimens were selected: Tinidazole , 2g twice daily for 14 days. At the same time, metronidazole, 400 mg, daily, vaginal administration for 14 days.
  Tinidazole , 1g three times daily for 14 days. At the same time, metronidazole, 400 mg, daily, vaginal administration for 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tinidazole 56 (Experimental): Tinidazole , 2g， twice daily for 14 days. At the same time, metronidazole, 400 mg, once a day, vaginal administration, 14 days.
  Interventions: Drug: Tinidazole 42
- Tinidazole 42 (Experimental): Tinidazole , 1g, three times daily for 14 days. At the same time, metronidazole, 400 mg, once a day, vaginal administration, 14 days.
  Interventions: Drug: Tinidazole 56

INTERVENTIONS:
Drug: Tinidazole 56 — Tinidazole , 2g， twice daily for 14 days. At the same time, metronidazole, 400 mg, once a day, vaginal administration, 14 days.
  Other Names: Tinidazole M56
  Arms: Tinidazole 42
Drug: Tinidazole 42 — Tinidazole , 1g, three times daily for 14 days. At the same time, metronidazole, 400 mg, once a day, vaginal administration, 14 days.
  Other Names: Tinidazole M42
  Arms: Tinidazole 56

SUMMARY:
We compare two oral tinidazole regimens for refractory trichomonas vaginitis.

DETAILED DESCRIPTION:
Refractory trichomonas vaginitis has become a clinical problem, which has a direct impact on the health and life of patients. Refractory trichomonas vaginitis is mainly caused by drug resistance of trichomonas. Drug resistant trichomonas has appeared China. Increasing the dosage of anti trichomonal drugs is the main treatment method at present. The aim of this study was to evaluate the efficacy and safety of two oral tinidazole regimens for refractory trichomonas vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* Women be at least 18 years of age
* Failure of conventional treatment (recommended by guidelines including tinidazole, 2g once daily for 5-7 days)

Exclusion Criteria:

* Allergy to metronidazole or tinidazol
* Pregnant or nursing
* HIV or other chronic disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Cure rate of refractory trichomoniasis | 24 weeks
  Evaluate the efficacy of oral tinidazole tablets in the treatment of refractory trichomoniasis.Diagnosis of vaginal trichomoniasis is performed by microscopy of vaginal secretions. Cure or failure was based on positive or negative T. vaginalis on vaginal secretions by microscopy examination.

SECONDARY OUTCOMES:
Safety of tinidazole tablets | 24 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. Test of blood routine,liver function, kidney function ,and urine routine will be done before treatment.The same test will be were reviewed within 1 week after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shangrong Fan Fan, M.D., Principal Investigator — Peking University Shenzhen Hospital
Locations (4):
- China (4):
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, School of Clinical Medicine, Tsinghua University, Beijing
  - Peking University First Hospital, Beijing